CLINICAL TRIAL: NCT04388293
Title: Using Antibiotics Wisely - Development of National Neonatal Intensive Care Unit-specific ASP
Brief Title: Using Antibiotics Wisely - An Antimicrobial Stewardship Program
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: University of Calgary (Other); University of Toronto (Other); Memorial University of Newfoundland (Other); Children's Hospital of Eastern Ontario (Other); Université de Montréal (Other)
Responsible Party: Principal Investigator, Joseph Ting, Principal Investigator, University of Alberta
Other Study IDs: H19-02490
Record Dates: First submitted 2020-05-10; First posted 2020-05-14 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Multi-Drug Resistant Organisms; Late-Onset Sepsis, Neonatal; Antimicrobial Resistance
Keywords: Antimicrobial Stewardship; Prematurity; Neonate
MeSH Terms: conditions — Neonatal Sepsis; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exposure of interest — Very Low Birth Weight infants admitted to tertiary NICUs in Canada.

SUMMARY:
There are significant variations in antimicrobial consumption across Canadian Neonatal Intensive Care Units (NICUs). Inappropriate and overuse of antibiotics can result in antimicrobial resistance and adverse outcomes among vulnerable neonatal populations. There are limited data on broad-spectrum antimicrobial use, multi-drug resistant organisms (MDRO) prevalence, and effective NICU-specific antimicrobial stewardship strategies. The aim of this study is to develop and implement NICU-specific antimicrobial stewardship strategies at both national and individual unit levels to promote optimal antimicrobial use and decrease the incidence of MDROs.

DETAILED DESCRIPTION:
Purpose: The investigators aim to develop and implement NICU-specific Antimicrobial Stewardship Program (ASP) strategies at both national and individual unit levels to promote optimal antimicrobial use and decrease the incidence of multi-drug resistant organisms (MDRO) in Canada.

Hypothesis: The investigators expect to find:

* Significant national variation in broad-spectrum antimicrobial use, which will not be correlated with rates of sepsis. High antimicrobial consumption rates may be associated with limited existing ASP resources and increased neonatal morbidity related to inflammatory cascades.
* Significant national variation in the prevalence of MDROs across NICUs.
* Differences in empirical antimicrobial regimens may be associated with MDRO prevalence, and the variation in antimicrobial use may explain some variation in neonatal morbidity.

Study Population and Sample Size: The study population will include very-low-birth-weight (VLBW) infants (i.e., the group of infants neonates with the highest risk of infections within NICUs) admitted to participating tertiary NICUs in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Very-low-birth-weight infants admitted to participating tertiary NICUs in Canada.

Exclusion Criteria:

* infants with major congenital anomalies

Ages: 22 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include all VLBW infants admitted to participating tertiary NICUs in Canada. The investigators will exclude infants with major congenital anomalies to avoid confounding factors when analyzing the impact of antimicrobial use and MDRO on neonatal outcomes. All VLBW infants will be included in the primary MDRO prevalence analysis. The investigators expect ~2000 VLBW infants with culture-proven infections in the study period.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Days of therapy/1000 patient-day of each category of antimicrobial consumption | 2020-2025
Prevalence of multi-drug resistant organisms in infections among very-low-birth-weight neonates during their NICU stay | 2020-2025

SECONDARY OUTCOMES:
Association between multi-drug resistant organisms, broad-spectrum antimicrobial use, neonatal outcomes and existing Antimicrobial Stewardship Programs & screening policies. | 2020-2025

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ting JY, Roberts A, Tilley P, Robinson JL, Dunn MS, Paquette V, Lee KS, Shah V, Yoon E, Richter LL, Lodha A, Shivananda S, Thampi N, Autmizguine J, Shah PS; Canadian Neonatal Network Investigators. Development of a national neonatal intensive care unit-specific antimicrobial stewardship programme in Canada: protocol for a cohort study. BMJ Open. 2020 Dec 10;10(12):e043403. doi: 10.1136/bmjopen-2020-043403. PMID 33303471